CLINICAL TRIAL: NCT01992679
Title: Body Weight Supported Treadmill Training in Advanced Multiple Sclerosis
Brief Title: Body Weight Supported Treadmill Training in Persons With Multiple Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Jacob Sosnoff, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMSS-IL-011
Record Dates: First submitted 2013-11-12; First posted 2013-11-25 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Participants in the control group will undergo the same assessments but receive no exercise stimulus and be asked to maintain current physical levels
- Exercise group (Experimental): The exercise program will consist of biweekly training sessions for 20 weeks. Per neurorecovery network guidelines, each training session will include a minimum of 20 minutes of locomotor training and 20 minutes of balance training.
  Interventions: Behavioral: Exercise group

INTERVENTIONS:
Behavioral: Exercise group — The BWSTT program will consist of biweekly training sessions for 20 weeks. Per neurorecovery network guidelines, each training session will include a minimum of 20 minutes of locomotor training and 20 minutes of balance training. Training will take place on a Therastride which consists of a treadmill with an air pressure powered pulley system connected to a harness system. The locomotor training strategy focuses on proper gait mechanics, including weight bearing, shifting and maintaining body positioning. Manipulating the participant's legs is done in such a way as to provide appropriate sensory-motor cues that facilitate the development and refinement of walking pattern.
  Other Names: Body-weight supported treadmill triaining
  Arms: Exercise group

SUMMARY:
There is growing evidence that exercise-based rehabilitation results in improvements in mobility and participation in persons with multiple sclerosis (MS). However, the vast majority of the scientific evidence in support of this view is based on persons with MS who have minimal mobility impairment. This is partially due to the lack of accessible exercise equipment and facilities available to persons with severe mobility limitations.

One option available to persons with severe mobility limitations is body weight supported treadmill training. Indeed, this rehabilitation approach has been utilized with some success in various clinical populations, such as stroke and spinal cord injury, and is believed to target neuroplasticity. Specific to persons with MS, body weight supported treadmill training has shown great promise in improving quality of life, symptoms and functional mobility in two small (n=4 and n=6) pilot investigations. However, previous research has been hampered by methodological limitations including small sample size, lack of a control group and limited training sessions. Consequently, no firm conclusion regarding the benefit of body weighted supported treadmill training in persons with MS can be drawn. The proposed project seeks to determine if twenty-weeks of body weight supported treadmill training leads to improvements in physiological function, mobility and quality of life in persons with MS with severe mobility limitations. The outcomes of this project have the potential to lead to new rehabilitation approaches capable of improving function and quality of life in persons with advanced MS.

DETAILED DESCRIPTION:
One option available to persons with severe mobility limitations is body weight supported treadmill training. Indeed, this rehabilitation approach has been utilized with some success in various clinical populations, such as stroke and spinal cord injury, and is believed to target neuroplasticity. Specific to persons with MS, body weight supported treadmill training has shown great promise in improving quality of life, symptoms and functional mobility in two small (n=4 and n=6) pilot investigations. However, previous research has been hampered by methodological limitations including small sample size, lack of a control group and limited training sessions. Consequently, no firm conclusion regarding the benefit of body weighted supported treadmill training in persons with MS can be drawn. The proposed project seeks to determine if twenty-weeks of body weight supported treadmill training leads to improvements in physiological function, mobility and quality of life in persons with MS with severe mobility limitations. The outcomes of this project have the potential to lead to new rehabilitation approaches capable of improving function and quality of life in persons with advanced MS.

ELIGIBILITY:
Inclusion Criteria:

* The criteria for inclusion are physician confirmed MS diagnosis, relapse free in the last 30 days, ability to voluntarily contract either quadriceps (e.g. extend their knee), willingness to complete 20 week intervention, and physician approval to engage in manual BWSTT. The diagnosis of MS based on either Poser's or McDonald's criteria and its type based on Lublin and Reingold criteria will be confirmed by the patient's neurologist using a standard form letter.

Exclusion Criteria:

* The criteria for exclusion are having a relapse in the last 30 days, inability to contract the quadriceps, and unwilling to complete the 20 week intervention.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Clinical Disability | 5 months
  Clinical disability will be indexed by expanded disability status scale.
Quality of Life | 5 months
  Quality of life will be indexed with the Multiple Sclerosis Quality of Life-54 (MSQoL-54) and participation will be indexed with the community participation indicator.

SECONDARY OUTCOMES:
Walking function | 5 months
  Walking speed will be quantified with the Timed 25-Foot Walk and walking endurance will be quantified with the 6-Minute Walk. The Multiple Sclerosis Walking Scale-12 (MSWS-12) will be used as a self-reported measure of walking impairment.
Balance | 5 months
  Balance will be quantified with the Berg Balance Scale (BBS); self-report of balance confidence (ABC), and force platform metrics (sway range and velocity).
Cardiorespiratory fitness | 5 months
  Cardiorespiratory fitness will be measured as peak oxygen consumption (VO2peak) using an incremental exercise test using an total body recumbent stepper and an open-circuit spirometry system.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Sosnoff, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois UC, Urbana-Champaign, Illinois, United States